CLINICAL TRIAL: NCT02673281
Title: Activation of Brain Centers Responsible for Decreasing Appetite and Improvement of the Cardiometabolic Profile by Short-term Walnut Consumption in Obesity: A Pilot Study
Brief Title: Activation of Brain Centers by Short-term Walnut Consumption in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christos Mantzoros, MD DSc h.c. PhD mult, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2015P000343
Record Dates: First submitted 2016-01-13; First posted 2016-02-03 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Obesity
Keywords: walnuts; brain; appetite; energy intake; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walnut shake (Experimental): All subjects will have 2 5-day visits to the BIDMC clinical research center, one where they will receive active milkshake containing 48g of walnuts daily in a single morning meal instead of breakfast, and another where they will receive a "placebo" milkshake without nuts
  Interventions: Other: Walnut shake
- Placebo shake (Placebo Comparator): All subjects will have 2 5-day visits to the BIDMC clinical research center, one where they will receive active milkshake containing 48g of walnuts daily in a single morning meal instead of breakfast, and another where they will receive a "placebo" milkshake without nuts
  Interventions: Other: Placebo shake

INTERVENTIONS:
Other: Walnut shake — walnut shake will be administered for 5 days as a morning snack instead of a typical breakfast
  Arms: Walnut shake
Other: Placebo shake — placebo shake will be administered for 5 days as a morning snack instead of a typical breakfast
  Arms: Placebo shake

SUMMARY:
The purposes of the study are:

* Study Aim 1. To assess the mechanisms underlying the biological effects of short-term walnut consumption on appetite with functional magnetic resonance imaging (fMRI) and assessing neurocognitive function/memory
* Study Aim 2. To investigate the effects of walnut consumption (48g per day over 5 days) on appetite and satiety by analyzing molecules which regulate energy homeostasis such as adipokines, as well as resting metabolic rate which measures energy expenditure.
* Study Aim 3. To investigate the effects of walnuts (48g per day over 5 days) on insulin resistance, lipids, and inflammatory markers in obesity as well as the effect of walnuts when consumed as part of a mixed meal, on glucose excursions, insulin secretion and the excretion of gut peptides and free fatty acids.

DETAILED DESCRIPTION:
Study Overview:

The study is a short-term, pilot, double-blinded, randomized, cross-over inpatient study testing the effects of either 48 g of walnuts per day vs. an ad libitum diet without walnuts on appetite and satiety, insulin resistance, basal metabolic rate, lipids, adipokines, heart rate, vascular reactivity, and markers of inflammation. The investigators propose that subjects stay in the controlled environment of our Clinical Research Center (CRC) for the entire duration of each arm of the study (5 days), which will be separated from the other arm by a one month long wash out period. Walnuts/placebo administration will be in the form of a milkshake with identical macronutrient content. Each study subject will be fed an identical diet during both admissions to minimize variability.

Study Design:

Screening: Potential subjects will be initially screened through telephone to determine that they are eligible for inclusion in the study according to the inclusion/exclusion criteria. If they pass the phone screening then they will be asked to come at CRC for a screening visit. They will have a detailed medical history, physical exam, fasting lab tests such as fructosamine, international normalized ratio (INR), prothrombin time (PT), complete blood count (CBC), metabolic panel including glucose and lipid profile, electrocardiogram (EKG), vitals, anthropometry and pregnancy test for women and if eligible for participation they will sign the informed consent of the study.

Subjects meeting eligibility criteria will be randomized to start with either the active intervention or placebo. Subjects will complete a 3-day food diary prior to visit 1 to document baseline diet. They will also meet the dietitian who will advise them on following a prudent diet and maintaining a stable exercise pattern for 2 weeks before the first visit and between both visits. Subjects will also be advised to avoid walnuts during this period. Subjects will also be required to maintain their weight +/- 3kg between screening and between study visits.

In-patient CRC Admission: In order to ensure stable study conditions, eligible subjects will be asked to stay in the CRC of the Beth Israel Deaconess Medical Center (BIDMC) for a period of 5 days on each of the study visits. They will receive advice on isocaloric diet but will be allowed to eat ad libitum and will be randomized prior to the first visit regarding the sequence of the study visits. All subjects will have 2 5-day visits to the CRC, one where they receive active milkshake containing 48g of walnuts daily in a single morning meal instead of breakfast, and another where they receive a "placebo" milkshake without nuts. Subjects will have their hunger assessed using visual analog scales before breakfast, lunch and dinner each day. These inpatient visits will be separated from each other by a 1-month washout period. Subjects and investigators will be blinded regarding the study sequence.

For each of the inpatient series, subjects will be admitted to CRC the night before the first day of the study. On day 1, subjects will have baseline measures such as vitals, anthropometry, brief medical history, physical exam, pregnancy test for women. Prior to leaving the CRC on day 5, subjects will again have vitals, blood draws for several markers including fructosamine, lipid panel, high sensitivity c-reactive protein (hsCRP), adiponectin and leptin, resting metabolic rate (RMR), anthropometry and body composition measures. On this last day, they will also undergo neurocognitive testing and an fMRI at the fasting state while viewing food cues and a mixed meal challenge either with or without walnuts. Subjects will be discharged from the CRC after their final testing and after evaluating the milkshake they were consuming on day 5 and will resume their normal diet for a period of 4 weeks after which time they will return to the CRC for a further 5 days for the second study visit. Prior Visit 2 participants will complete another 3-day food diary. If they received placebo milkshake on the first visit, they will have the walnut milkshake on the second visit and vice-versa.

ELIGIBILITY:
Inclusion Criteria:

* 10 otherwise healthy men or women, 18-65 years old, with a Body Mass Index (BMI) >30kg/m2 or a BMI >27kg/m2 with comorbidities that would require treatment for obesity (assessed through the screening questionnaire and the medical history and physical exam examination during the screening visit).

Exclusion Criteria:

* Diagnosis of diabetes, defined per American Diabetes Association (ADA) criteria as hemoglobin a1c (Hba1c) > 7.0% and/or fasting glucose > 125 mg/dL and/or random glucose > 200 mg/dL
* Subjects with any medical condition or on any treatment which would interfere with the study outcomes or would make participation potentially harmful such as pregnancy or breastfeeding, anemia, unstable heart disease, stroke, malabsorption syndromes according to a detailed medical history.
* Present alcoholism or drug abuse or use of any medications the dose of which would be changing or plan to initiate any new medications during the study period. These conditions will be screened for by a detailed history and systems review.
* Individuals with nut allergies or allergies to the ingredients of the milkshake (walnuts, mangos, strawberries, bananas, berry medley, pineapple juice, safflower oil, walnut flavoring) are excluded.
* Subjects with any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g. cochlear implants, pacemakers, neuron or biostimulators, electronic infusion pumps, etc.)
* Subjects with any type of metallic implant that could potentially be displaced or damaged during MRI, such as aneurysm clips, metallic skull plates, surgical implants etc. or metal containing tattoos.
* Anxiety of small spaces and/or claustrophobia
* Subjects with neurological or psychiatric problems which may interfere with or complicate testing (e.g. presence of titubation)
* Body weight above the limitation of the MRI scanning table (330lbs/150 Kg) or body dimensions that could difficult the performance of the scan.
* Subjects who cannot adhere to the experimental protocol for any reason
* Uncontrolled infectious diseases (e.g. human immunodeficiency virus (HIV), hepatitis, chronic infections etc)
* Any uncontrolled endocrine condition, e.g. Cushing's, Acromegaly, etc
* Any cancers or lymphoma
* Eating disorders like anorexia, bulimia
* Weight loss surgery or gastrectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
brain centers activation related to food intake assessed using functional magnetic resonance imaging (fMRI) | fasting Day 5
  The investigators will use functional magnetic resonance imaging (fMRI) to identify brain centers activation related to food intake after the consumption of the walnut shake compared to the placebo shake.

CONTACTS AND LOCATIONS:
Overall Officials: Christos S Mantzoros, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Clinical Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant data will be kept confidential.

REFERENCES:
- [Derived] Tuccinardi D, Perakakis N, Farr OM, Upadhyay J, Mantzoros CS. Branched-Chain Amino Acids in relation to food preferences and insulin resistance in obese subjects consuming walnuts: A cross-over, randomized, double-blind, placebo-controlled inpatient physiology study. Clin Nutr. 2021 May;40(5):3032-3036. doi: 10.1016/j.clnu.2021.01.020. Epub 2021 Jan 23. PMID 33541836
- [Derived] Farr OM, Tuccinardi D, Upadhyay J, Oussaada SM, Mantzoros CS. Walnut consumption increases activation of the insula to highly desirable food cues: A randomized, double-blind, placebo-controlled, cross-over fMRI study. Diabetes Obes Metab. 2018 Jan;20(1):173-177. doi: 10.1111/dom.13060. Epub 2017 Aug 17. PMID 28715141